CLINICAL TRIAL: NCT02618681
Title: Earlobe Creases Predict Prognosis in Chinese Patients With Acute Myocardial Infarction
Acronym: ELC-CHN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jing Qi (Other)
Responsible Party: Sponsor-Investigator, Jing Qi, Principal investigator, Liaoning University of Traditional Chinese Medicine
Organization: Liaoning University of Traditional Chinese Medicine (Other)
Other Study IDs: JQi
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Ear Abnormalities; Prognosis
Keywords: earlobe crease; acute myocardial infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AMI with earlobe crease: To observe the prognosis for AMI with earlobe crease
- AMI without earlobe crease: To observe the prognosis for AMI without earlobe crease

INTERVENTIONS:
Other:

SUMMARY:
To investigate the feasibility of the earlobe crease as an early prognostic predictor for acute myocardial infarction(AMI) in Chinese population.

DETAILED DESCRIPTION:
Primary Objective : 1 year primary composite end point (including the whole death, recurrent myocardial infarction, stroke, target vessel revascularization, stent thrombosis) in AMI patients with different types of earlobe crease.

Secondary objective:

1. The incidence of complications during hospitalization
2. The rate of rehospitalization due to cardiovascular disease
3. The incidence of revascularization at 1 year after AMI

ELIGIBILITY:
Inclusion Criteria:

1. Initial acute myocardial infarction(AMI)
2. Detection of a rise and/or fall of cardiac biomarker values (preferably cardiac troponin (cTn) with at least one value above the 99th percentile upper reference limit (URL)) and with at least one of the following:

   * Symptoms of ischemia
   * Development of pathologic Q waves in the electrocardiogram (ECG)
   * New or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB).
   * Identification of an intracoronary thrombus by angiography or autopsy
   * Imaging evidence of new loss of viable myocardium or a new regional wall motion abnormality.
3. Type 1 (spontaneous myocardial infarction(MI)) in the third universal definition of MI: MI consequent to a pathologic process in the wall of the coronary artery (eg, plaque erosion/rupture, fissuring, or dissection), resulting in intraluminal thrombus.
4. Infarct related artery (IRA) showed that acute thrombus formation, IRA occlusion or stenosis ≥95%、≥90%～95%、≤90%，thrombolysis in myocardial infarction (TIMI)0-3 flow.
5. PCI(percutaneous coronary intervention)intervention（PCI for STEMI within 12 hours after symptom onset）.
6. Signed informed consent.

Exclusion Criteria:

1. Combined valvular heart disease, cardiomyopathy, blood diseases, skin diseases, rheumatic diseases, ischemic cerebrovascular disease, tumor, etc.
2. Previous myocardial infarction.
3. Previous PCI and coronary artery bypass graft(CABG).
4. Chronic total occlusion(CTO)lesions.
5. Ear malformation.
6. Ocular diseases.
7. Participating in a clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute myocardial infarction
Sampling Method: Probability Sample
Enrollment: 902 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
primary composite end point (including the whole death, recurrent myocardial infarction, stroke, target vessel revascularization, stent thrombosis) in AMI patients with different types of earlobe crease. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Junwen Jiang, Doctor, Study Director — Liaoning University of Traditional Chinese Medecine
Locations (1):
- Jing, Shenyang, Liaoning, China